CLINICAL TRIAL: NCT03136276
Title: One Year Clinical Evaluation of IPS Empress CAD Versus Polished Celtra Duo Ceramic Laminate Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hayat Ibrahim Mahrous Ibrahim, assisstant lecturer, fixed prosthodontic department, faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19786
Record Dates: First submitted 2017-04-10; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Tooth Discoloration; Tooth Fractures; Diastema
MeSH Terms: conditions — Tooth Discoloration; Tooth Fractures; Diastema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPS Empress CAD (Active Comparator): Leucite Based glass Ceramics which is etchable ceramics and proved to have good success rate if used for laminate veneers
  Interventions: Other: IPS Empress CAD
- polished Celtra Duo (Experimental): Zirconia reinforced lithium silicate, it is a recent material with glass ceramics enriched with 10% zirconia that offers high strength properties
  Interventions: Other: polished Celtra Duo

INTERVENTIONS:
Other: IPS Empress CAD — standard etchable glass ceramics
  Other Names: leucite based glass ceramics
  Arms: IPS Empress CAD
Other: polished Celtra Duo — new glass ceramic material
  Other Names: zirconia reinforced lithium silicate (ZLS)
  Arms: polished Celtra Duo

SUMMARY:
When restoring teeth with IPS Empress laminate veneers, fracture of restorations may occur. So, material with higher mechanical properties is required. Celtra Duo is a new material with glass ceramics infiltrated by 10% zirconia particles which increase the fracture resistance of the material.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to be:

1. From 18-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations
3. Psychologically and physically able to tolerate conventional dental procedures
4. Patients with teeth problems indicated for laminate veneer:

   1. Discoloration
   2. Fracture not involving more than 50% enamel loss
   3. Mild malposition
   4. Diastema
   5. Enamel fluorosis
   6. Stained or defective restorations
5. Able to return for follow-up examinations and evaluation

Exclusion Criteria:

1. Patient with post and core endodontically treated teeth
2. Patient with fractured teeth of more than 50% enamel loss
3. Patients with poor oral hygiene and motivation
4. Pregnant women's
5. Patients in the growth stage with partially erupted teeth
6. Psychiatric problems or unrealistic expectations
7. Lack of opposing dentition in the area of interest
8. Patients involved in contact sports
9. Teeth with deep discoloration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Fracture | 1 year
  number of fractured laminates

IPD SHARING:
Plan to Share IPD: Undecided